CLINICAL TRIAL: NCT03265795
Title: Validity of PEEK PSI Containing Autogenous Bone Graft for Maxillary Reconstruction Following Lesion Enucleation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Zain, internal resident at oral and maxillofacial department, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: maxillary reconstruction
Record Dates: First submitted 2017-08-27; First posted 2017-08-29 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Maxillary Cyst

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEEK patient specific implant (Experimental): this PEEK (poly ether ether ketone) Patient Specific Implant containing autogenous bone graft is used in reconstruction of the bone and the original volume of maxillary sinus accurately (in terms of clinical and radiographic parameters).
  Interventions: Device: Poly Ether Ether Ketone PSI (patient specific implant).

INTERVENTIONS:
Device: Poly Ether Ether Ketone PSI (patient specific implant). — reconstruction of the bone and the original volume of maxillary sinus accurately (in terms of clinical and radiographic parameters).

SUMMARY:
Surgical ablation of large maxillary cysts usually results in considerable hard and soft tissue deficits that ultimately affect the final esthetic and functional outcomes. Reconstruction of such defects; whether primarily or secondarily; offers much better long-term outcomes. However, primary bony reconstruction becomes potentially complicated in many cases of such large cysts encroaching or involving the maxillary sinus where a communication with the maxillary sinus lining may be unavoidable.

Reconstruction of such defects can be accomplished using either vascularized or; more commonly; non-vascularized autogenous bone grafts. Different bone substitutes remain to be another viable option. The simultaneous use of titanium meshes provides physical three-dimensional support for the bone graft contained within as well as the overlying soft tissues. However, the drawbacks of titanium meshes in such defects remain to be mainly the difficulty in adequately shaping the mesh and the lack of proper isolation of the mesh contents from the maxillary sinus cavity.

ELIGIBILITY:
Inclusion Criteria:

1. Age of patients from 15 to 60 years old.
2. Patients with unilateral maxillary lesion encroaching maxillary sinus.
3. Dentulous or edentulous patients.
4. Patients should be free from any systemic disease that may affect normal healing of bone and predictable outcome.

Exclusion Criteria:

1. Patients with systemic diseases as history of radiation therapy or chemotherapy, hematological disorders, neuromotor disorders and autoimmune diseases (may affect normal healing).
2. Patients with bilateral maxillary lesions.
3. Children under 15 years old.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
oral health related quality of life | 4 months
  OHIP-49 questionaire

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gellrich NC, Schramm A, Hammer B, Rojas S, Cufi D, Lagreze W, Schmelzeisen R. Computer-assisted secondary reconstruction of unilateral posttraumatic orbital deformity. Plast Reconstr Surg. 2002 Nov;110(6):1417-29. doi: 10.1097/01.PRS.0000029807.35391.E5. PMID 12409759
- [Background] Eckardt A, Swennen GR. Virtual planning of composite mandibular reconstruction with free fibula bone graft. J Craniofac Surg. 2005 Nov;16(6):1137-40. doi: 10.1097/01.scs.0000186306.32042.96. PMID 16327572
- [Background] Lethaus B, Kessler P, Boeckman R, Poort LJ, Tolba R. Reconstruction of a maxillary defect with a fibula graft and titanium mesh using CAD/CAM techniques. Head Face Med. 2010 Jul 19;6:16. doi: 10.1186/1746-160X-6-16. PMID 20642821